CLINICAL TRIAL: NCT05213091
Title: The Effect of Otago Exercises on Fear of Falling, Balance, Empowerment and Functional Mobility in Elderly: A Randomized Controlled Trial
Brief Title: The Effect of Otago Exercises in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Naile Bilgili, Professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2021-465
Record Dates: First submitted 2021-12-24; First posted 2022-01-28 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Healthy Aging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research data/output measurements, analysis and reporting
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago Exercise Group (Experimental): Otago Exercise program wil be applied to the elderly.
  Interventions: Other: Otago Exercise Programme
- Control Group (No Intervention): The elderly wil be expected to continue their daily life.

INTERVENTIONS:
Other: Otago Exercise Programme — The first four weeks will be Otago Exercise Programme training and practice. For the next weeks, there will be institution visits and telephone interviews. Individuals will be given an Otago Exercise Programme training booklet, exercise chart and exercise diary to better manage this process. The research will be conducted in small groups (average 6-8).
  Other Names: Otago exercise programme training and implementation, phone call, institution visit
  Arms: Otago Exercise Group

SUMMARY:
Home-based and individually designed exercise program; It consists of warming up, strengthening, balance exercises and walking plan. The number, intensity and duration of the movements are personalized according to preference and ability and are progressed gradually. Elderly individuals are expected to do this set of exercises three times a week and walk for 30 minutes twice a week. Since the Otago Exercise Programme includes combined exercises, the outputs of the effectiveness of the program will be different. For this purpose, the effect of otago exercises on fear of falling, balance, strengthening and functional mobility will be determined in the elderly living in nursing homes.

DETAILED DESCRIPTION:
The first four weeks will be Otago Exercise Programme training and practice. For the next weeks, there will be institution visits and telephone interviews. Individuals will be given an Otago Exercise Programme training booklet, exercise chart and exercise diary to better manage this process. The research will be conducted in small groups (average 6-8). The control group is expected to continue their daily life. No attempt will be made by the researcher during the research process. Stratified randomization method according to age and gender was used in the study. The website was used to assign individuals meeting the inclusion criteria in each stratum to a determined number of groups. Masking will be done in terms of research data/output measurements (evaluator), statistician and reporting.

ELIGIBILITY:
Inclusion Criteria:

* To be 65 years or older
* To be literate
* Having no problem in verbal communication
* Not having a disability based on sight, hearing and lack of limbs
* Obtaining at least 91 points or more according to the Barthel Activities of Daily Living Index (to be mildly dependent or completely independent)
* Mini Mental Test to be 24 points and above
* Having a doctor's report that it will not interfere with exercise

Exclusion Criteria:

* Having a medical contraindication for exercise
* Having acute or terminal illnesses and serious chronic illnesses that limit participation in exercise sessions
* Having a lower extremity fracture in the past year
* Having had an operation in the last month
* Being diagnosed with any neuropsychiatric disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Modified Fall Efficacy Scale | Totally 12 weeks
  The scale is used to determine the possible fear of falling in elderly individuals. It is a visual analog scale consisting of fourteen questions. Items are scored from zero to ten (never safe=0, totally safe=10). A high score means high fall safety and proficiency.
Berg Balance Scale | Totally 12 weeks
  The scale was developed to evaluate the balance levels of elderly individuals. This scale consists of 14 items and each section is scored between 0 (bad) and 4 (best). The scale score is in the range of 0-56 points, and an increase in the score indicates that the balance is good. According to the total score obtained, "0-20 points: high risk of falling, balance disorder", "21-40 points: moderate risk of falling, presence of acceptable balance", "41-56 points: low risk of falling, presence of good balance" evaluated as ".
Elderly Empowerment Scale | Totally 12 weeks
  The scale is a short and practical tool for assessing the empowerment levels of the elderly. The scale, which consists of a total of eight questions and a single factor, is in the five-point Likert type. The lowest score obtained from the scale is 8, the highest score is 40.
30-Second Chair Stand Test | Totally 12 weeks
  It is a test that evaluates the sit-to-stand activity, lower extremity strength and dynamic balance of the individual. The number of times an individual sits and stands in 30 seconds is recorded. Three measurements will be made by giving rest intervals and the average will be recorded.
Handgrip Strength Measurement Test | Totally 12 weeks
  The purpose of the test is to test the maximum isometric contraction strength of the forearm muscles. The average of the three measurements will be taken and recorded.
Timed Up & Go | Totally 12 weeks
  It is a test that evaluates mobility and fall risk in elderly individuals. The individual is observed while getting up from the chair, walking 3 meters, turning, walking back and sitting again, and the elapsed time is recorded. If the elderly person completes this test in more than 12 seconds, it is considered as "at risk of falling". Three measurements will be made by giving rest intervals and the average will be taken.
6-Minute Walk Test | Totally 12 weeks
  It was developed to measure the functional capacity of individuals. In the six-minute walking test, the patient walks along a 30-meter straight corridor as fast as he can, but without running. How many meters he walked is measured and recorded. Three measurements will be made by giving rest intervals and the average will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Çankaya/Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No